CLINICAL TRIAL: NCT01013012
Title: Efficacy of Dexamethasone Added to Ramosetron for Preventing Postoperative Nausea and Vomiting in Highly Susceptible Patients Following Spine Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2007-0388
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Nausea; Vomiting
Keywords: highly susceptible patients following spine surgery
MeSH Terms: conditions — Nausea; Vomiting | interventions — ramosetron; Sodium Chloride; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): Group A : saline 1 ml + ramosetron 6μg/kg
  Interventions: Drug: ramosetron with saline
- Group B (Experimental): Group B : dexamethasone 4 mg + ramosetron 6μg/kg
  Interventions: Drug: ramosetron with dexamethasone

INTERVENTIONS:
Drug: ramosetron with saline — Group A : saline 1 ml, ramosetron 6μg/kg
  Arms: Group A
Drug: ramosetron with dexamethasone — Group B : dexamethasone 4 mg, ramosetron 6μg/kg
  Arms: Group B

SUMMARY:
The purpose of this study is to study the efficacy of dexamethasone added to ramosetron for preventing postoperative nausea and vomiting in highly susceptible patients following spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Ages 18 to 65 years old

Exclusion Criteria:

* Patients who is taking steroid or who had been treated for the gastrointestinal disease
* Patients who have troubles with the kidney or liver
* Patients transferring to the ICU after the surgery
* overfat patients
* Patients who had taken antiemetics within 24 hours before the surgery

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
the incidence of postoperative nausea and vomiting(PONV) | After spinal surgery
  incidence of overall postoperative nausea and vomiting (PONV) between combination of ramosetron and dexamethasone and ramosetron alone in highly susceptible patients